CLINICAL TRIAL: NCT00851240
Title: A Multiple Ascending Dose Study to Assess the Safety and Pharmacokinetics of Repeated Intravenous Doses of BTT-1023 in Patients With Rheumatoid Arthritis - a Double-blind Randomized Placebo-controlled Sequential Group Trial
Brief Title: BTT-1023 in Rheumatoid Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biotie Therapies Corp. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BTT12-CD015
Record Dates: First submitted 2009-02-02; First posted 2009-02-25 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; safety
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — timolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- BTT1023 (Experimental)
  Interventions: Drug: BTT-1023
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BTT-1023 — intravenous
  Arms: BTT1023
Drug: Placebo — Intravenous
  Arms: Placebo

SUMMARY:
Patients with adult-onset rheumatoid arthritis will be enrolled. They will be dosed with repeated intravenous doses of BTT-1023 or placebo. During the trial, the safety of the treatments and the pharmacokinetics of BTT-1023 will be assessed. The patient allocation to treatment groups will occur at random, and the actual treatment will not be revealed to the investigator or to the patient during the trial.

ELIGIBILITY:
Inclusion Criteria:

* adult-onset rheumatoid arthritis

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-02; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Incidence and intensity of adverse events | 17 wk

SECONDARY OUTCOMES:
Serum concentrations of the verum | 17 wk
Disease activity | 17 wk

CONTACTS AND LOCATIONS:
Overall Officials: Antero Kallio, MD, Study Director — Biotie Therapies Corp.
Locations (1):
- Sofia, Bulgaria, Sofia, Bulgaria